CLINICAL TRIAL: NCT04847245
Title: A Randomized Controlled, Single-blind, Esketamine Adjuvant Therapy for the Efficacy and Safety of Patients With Chronic Visceral Pain Comorbid Major Depressive Disorder
Brief Title: Esketamine Adjuvant Therapy for Patients With Chronic Visceral Pain Comorbid Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Si Tianmei, Professor, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Esketamine20210221
Record Dates: First submitted 2021-03-14; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Chronic Visceral Pain; Major Depressive Disorder
Keywords: Esketamine; Pregabalin; Efficacy and Safety; Chronic Visceral Pain; Major depressive disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Pregabalin; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pregabalin group (Active Comparator): Pregabalin capsules were administered orally (75 mg, tid), combined administration of duloxetine.
  Interventions: Drug: Pregabalin 75mg tid + Duloxetine
- 0.125 mg/kg esketamine group (Experimental): Intravenous administration of esketamine 0.125 mg/kg，and duloxetine is co- administered orally.
  Interventions: Drug: Intravenous administration of esketamine 0.125 mg/kg+Duloxetine
- 0.25 mg/kg esketamine group (Experimental): Intravenous administration of esketamine 0.25mg/kg，and duloxetine is co- administered orally.
  Interventions: Drug: Intravenous administration of esketamine 0.25 mg/kg +Duloxetine
- 0.50 mg/kg esketamine group (Experimental): Intravenous administration of esketamine 0.50 mg/kg，and duloxetine is co- administered orally.
  Interventions: Drug: Intravenous administration of esketamine 0.50 mg/kg+Duloxetine

INTERVENTIONS:
Drug: Pregabalin 75mg tid + Duloxetine — Pregabalin capsules were administered orally (75 mg, 3 times a day), combined administration of duloxetine (60-120 mg/day）.
  Arms: Pregabalin group
Drug: Intravenous administration of esketamine 0.125 mg/kg+Duloxetine — Intravenous administration of esketamine 0.125 mg/kg （2 times per week)， combined oral administration of duloxetine (60-120 mg/day）
  Arms: 0.125 mg/kg esketamine group
Drug: Intravenous administration of esketamine 0.25 mg/kg +Duloxetine — Intravenous administration of esketamine 0.25 mg/kg （2 times per week)， combined oral administration of duloxetine (60-120 mg/day）
  Arms: 0.25 mg/kg esketamine group
Drug: Intravenous administration of esketamine 0.50 mg/kg+Duloxetine — Intravenous administration of esketamine 0.50 mg/kg （2 times per week)， combined oral administration of duloxetine (60-120 mg/day）
  Arms: 0.50 mg/kg esketamine group

SUMMARY:
Ketamine is a dissociative anesthetic and powerful analgesic. At low doses, ketamine can desensitize the central pain pathway and modulate opioid receptors. Studies have generally found that preoperative use of ketamine can reduce opioid consumption by approximately 50% and sub-anaesthetic doses of it have a rapid antidepressant effect, especially refractory depression. Studies have confirmed that esketamine, the S(+) enantiomer of ketamine, has a stronger affinity for NMDA receptors, which can achieve the same effect at smaller doses. While the incidence of neuropsychiatric side effects is significantly lower. On March 4, 2019, the U.S. Food and Drug Administration (FDA) first approved esketamine nasal spray with a new mechanism of action for the treatment of adult patients with refractory depression. Based on the analgesic and antidepressant effects of ketamine, the investigators speculate that esketamine may be effective for patients with chronic visceral pain comorbid depression. At present, the research evidence in this area is relatively lacking. Therefore, this study aims to explore the difference in the efficacy and safety of esketamine as an adjuvant therapy and positive control drug-pregabalin in patients with chronic visceral pain comorbid depression.

Detailed Description: According to the inclusion criteria and exclusion criteria, select patients with chronic visceral pain comorbid depression.

Filtering and grouping period: During this phase, the patient will sign an informed consent form, and then conduct a structured clinical evaluation to determine whether it meets the "depressive disorder" in the DSM-IV-TR diagnostic criteria. According to the ICD-11, determine whether the patients have chronic visceral pain.

Acute treatment period: Randomize patients into the following treatment groups: intravenous administration of esketamine (3 groups, 0.125, 0.25, 0.50 mg/kg)， and duloxetine is co- administered orally. Pregabalin capsules were administered combined with duloxetine orally.

observation period: After 2 weeks, esketamine treatment was discontinued, and observation was continued for 2 weeks. Maintain duloxetine and pregabalin treatment.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 to 55
2. Those who can understand and obey the research plan
3. Sign the informed consent form voluntarily
4. Those who meet the DSM-IV-TR depression diagnostic criteria and have first or second episodes of depression
5. Hamilton Depression Scale score ≥ 14 points
6. Those who meet the ICD-11 pain diagnostic criteria, and visual analogue scale score ≥ 7 points. Those who have chronic visceral pain instead of cancer pain.
7. No systemic use of antidepressants and analgesics within 2 weeks after enrollment.

   -

Exclusion Criteria:

1. Female patients who are pregnant, breastfeeding, or preparing to conceive
2. Allergic to duloxetine or pregabalin in the past.
3. A history of serious or unstable physical diseases, such as cardiovascular/liver/kidney/respiratory/ endocrine/nervous/ blood system disease.
4. A history of epileptic seizures or brain injury, or any neurological disease (including multiple sclerosis, degenerative diseases such as acute lateral sclerosis, Parkinson's disease and movement disorders, etc.);
5. In the last 12 months, the patient has the following medical history or its main diagnosis (DSM-IV-TR) is organic mental disorder, schizophrenia, schizoaffective mental disorder, delusional mental disorder, indeterminate mental disorder, Bipolar disorder, psychotic characteristics that are coordinated or uncoordinated with the mood, and history of substance abuse (including alcohol, psychoactive substances, etc.).
6. Patients with a history of adverse reactions to multiple drugs.
7. The patient is taking psychotropic drugs, including benzodiazepines, sleeping pills, anticonvulsants, etc.
8. During the depressive episode, treatment with at least 2 antidepressants in a sufficient course of treatment or at least one SSRI antidepressant treatment is ineffective. A sufficient dose of treatment means treatment with fluoxetine ≥40 mg/day (or sertraline ≥100 mg/day, paroxetine> 40 mg/day, fluvoxamine> 100 mg/day, citalopram> 40 mg /Day, escitalopram> 20 mg/day, venlafaxine> 150 mg/day, duloxetine> 80 mg/day)
9. Received electroconvulsive therapy within 6 months before enrollment.
10. Those who are currently at serious risk of suicide, and a score of 3 or higher in item 3 of the 17-HAMD .

    -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Day 0 to Day 28
  The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations, including those with chronic visceral pain. The minimus value is 0 and the maximum value is 10. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (HAMD) | Day 0 to Day 28
  The questionnaire is designed for adults and is used to rate the severity of their depression by probing mood, feelings of guilt, suicide ideation, insomnia, agitation or retardation, anxiety, weight loss, and somatic symptoms. The minimum value is 0 and the maximum value is 52. Higher scores mean a worse outcome.
Short Form 12 Health Survey (SF-12) | Day 0 to Day 28
  SF-12 is a 12-item, patient-reported survey of patient health, and is widely used since it produces similar results for physical and mental health scores with far less respondent burden for producing scores of overall mental and physical well-being. The SF-12 yields an eight-scale profile of scores as well as physical and mental health summary measures. Answers to questions of these subscales are combined (weighted) with Physical Component Summary (PCS-12) and Mental Component Summary (MCS-12) scale scores. SF-12 scales and summary measures are scored so that a higher score indicates a better health state. After recoding raw scores for some items (BP, GH, VT, and one item from MH), the raw scores could be transformed to provide scores for eight scales, each ranging from 0 (the worst) to 100 (the best).
Hamilton Anxiety Scale (HAMA) | Day 0 to Day 28
  The HAMA is a psychological questionnaire used by clinicians to rate the severity of a patient's anxiety. The scale consists of 14 items designed to assess the severity of a patient's anxiety. Each of the 14 items contains a number of symptoms, and each group of symptoms is rated on a scale of zero to four, with four being the most severe. The minimum value is 0 and the maximum value is 56. Higher scores mean a worse outcome.
Changes in serum inflammatory factors | Day 0 to Day 28
  Explore the action mechanism of esketamine on patients with chronic visceral pain comorbid depression from the level of blood inflammatory factors, including cytokines IL-1beta, IL-6, IL-8, IL-10, IL-12p70, TNF-alpha, etc.
Electroencephalogram (EEG) | Day 0 to Day 28
  Calculate the time-frequency characteristics of EEG data in each frequency band (delta wave, <4 Hz; theta wave, 4-8 Hz; alpha wave, 8-12 Hz and beta wave, 12-30 Hz) during the study period.
Functional magnetic resonance imaging (fMRI) | Day 0 to Day 28
  The regional brain activity, including fractional amplitude of low frequency fluctuation (fALFF) and regional homogeneity (ReHo) values, will be computed and assessed. In addtion, the large-scale brain networks and edge-wise connections in patients will be explored based on the theory of brain networks during the study period.